CLINICAL TRIAL: NCT06499896
Title: Phase II Trial of Healthy-donor Derived Full-spectrum Microbiome Therapeutic MTP-101-C in Steroid Relapse/Refractory Immune-related Cutaneous Adverse Events (irCAEs) and Immune-mediated Colitis (IMC) (FMT-ELIMINATE)
Brief Title: Healthy-donor Microbiome MTP-101-C in Steroid Relapse/Refractory Immune-related Cutaneous Adverse Events (irCAEs) and Immune-mediated Colitis (IMC)
Acronym: FMT-ELIMINATE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Diwakar Davar (Other)
Collaborators: Stanley Marks Fund for Cancer Research (Unknown); Cures Within Reach (Other)
Responsible Party: Sponsor-Investigator, Diwakar Davar, Assistant Professor of Medical oncology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCC 23-158
Record Dates: First submitted 2024-07-01; First posted 2024-07-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Immune-mediated Colitis (IMC); Immune-related Dermatitis
Keywords: gut microbiome; anti-PD-1 therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MTP-101-C (Cohort 1: Steroid R/R biologic-naive dermatitis) (Experimental): Patients given MTP-101-C (encapsulated fecal microbiota, containing ~5 x 1011 bacteria derived from healthy donors).
  Dosing:
  5 capsules/day (Day 1); 2 capsules/day (D2-D28)
  Interventions: Biological: MTP-101-C
- MTP-101-C (Cohort 2: Steroid R/R biologic-naive colitis) (Experimental): Patients given MTP-101-C (encapsulated fecal microbiota, containing ~5 x 1011 bacteria derived from healthy donors).
  Dosing:
  5 capsules/day (Day 1); 2 capsules/day (D2-D28)
  Interventions: Biological: MTP-101-C

INTERVENTIONS:
Biological: MTP-101-C — MTP-101-C is a screened, freeze-dried, encapsulated, full spectrum, healthy donor fecal microbiota product.

SUMMARY:
Multiple retrospective studies suggest that the administration of corticosteroids to treat irAEs is safe, and does not compromise efficacy of ICI therapy in cancer patients. While ~67% of patients respond to corticosteroids, 33% of patients require biologic therapy such as TNFα inhibitors (e.g. infliximab), integrin α4β7 inhibitors (e.g. vedolizumab), or JAK/STAT inhibitors (e.g. tofactinib). This study aims to determine that distinct pathobionts govern the development of irCAE and IMC; and that the administration of hdFMT may reverse steroid-refractory irCAEs or IMC. The use of hdFMT has been shown to be effective in steroid and biologic (TNFα and/or integrin α₄β₇ inhibitor) refractory colitis in PD-1 and/or CTLA-4 ICI treated cancer patients in single-institution case series.

DETAILED DESCRIPTION:
The study will be conducted over a 42-day period. Patients receiving anti-PD(L)1 and/or anti-CTLA-4 singly or in combination with other investigational agents are eligible to enroll. Enrollment is not limited by setting (adjuvant, metastatic) and/or line of therapy (1L, 2L etc.). Once enrolled, patients will be enrolled to receive MTP-101-C (encapsulated fecal microbiota, containing ~5 x 1011 bacteria derived from healthy donors) without prior antibiotic conditioning. MTP-101-C will be continued for 28 days during which steroids will be tapered rapidly. irAE endpoint assessment will be repeated following completion of hdFMT (D+28 to D+35) and at 6 weeks (D+42 to D+49). Biospecimens will be obtained periodically. The total duration of MTP-101-C therapy is 4 weeks. This study aims to determine distinct pathobionts govern the development of distinct irAEs including steroid-refractory irCAE or IMC; and that the administration of hdFMT ameliorates irCAE or IMC based on validated cohort-specific assessments: modified CTCAE grading system (cohort 1) or endoscopic assessment scale (full Mayo score, FMS) (cohort 2). Further, this trial aims to show that amelioration of inflammatory pathology is associated with key secondary objectives including: 1) improvements in an irAE toxicity-specific PRO FACT-ICM; and 2) clinically assessment scales. Also, this study will measure the correlation between symptom amelioration and changes in integrated biomarkers include measures of intestinal inflammation (fecal calprotectin), bacterial engraftment (metagenomic) and reactivity to donor bacteria (IgG-seq); exploring the effects of microbiome modulation upon time to steroid discontinuation, time to resumption of therapy, time to next treatment clinical remission by FMS, clinical remission by PMS, and key survival endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Able to swallow oral medication.
* The participant provides written informed consent for the trial.
* Willingness to use contraception for duration of trial participation. Male participants: A male participant must agree to use a contraception per protocol during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period.

Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

Not a woman of childbearing potential (WOCBP) per protocol; OR A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.

-Clinically confirmed inflammatory irCAE or endoscopically confirmed IMC. Cohort 1 (irCAE): Patients with maculopapular rash, psoriasiform, lichenoid eruptions or bullous pemphigoid of at least grade 3 severity per CTCAE grading system (i.e. >30% BSA with moderate or severe symptoms) during Screening.

Cohort 2 (IMC): Endoscopically confirmed inflammatory colitis as determined by colonoscopy or flexible sigmoidoscopy during Screening with minimum severity per Mayo endoscopic subscore 1-¬3 [MES1-3].

-Prior receipt of anti-PD(L)1 and/or anti-CTLA-4 singly or in combination with other approved or investigational agents including chemotherapy or targeted therapy.

NOTE: Patient may have received or are receiving ICI therapy as standard-of-care or part of a clinical trial.

Patient must have received treatment with an anti-PD-(L)1 ICI, anti-CTLA-4 ICI singly and/or in combination with other approved and/or investigational anti-cancer agent(s), as their most recent therapy prior to development of colitis.

Cohort 1 (steroid relapsed/refractory Grade ≥3 irCAE) only

* Receipt of high-dose systemic corticosteroids defined as 1-2mg/kg prednisone equivalent daily (either oral or intravenous) with a taper over 4-6 weeks as defined by society consensus guidelines102-105; AND
* No receipt of biologic such as but not limited to (dupilumab, rituximab) prior to enrollment.
* NOTE: Patients must have received steroids to be eligible.
* NOTE: Steroid "resistant" disease: patients whose symptoms responded (reduction in a CTCAE grade) initially but who developed recurrence upon steroid taper or discontinuation.
* NOTE: Steroid "refractory" disease: patients whose symptoms have not clinically improved by a CTCAE grade in ≥48 hours or maximum of 14 days.

Cohort 2 (steroid-relapsed/refractory Grade ≥3 IMC) only

* Receipt of high-dose systemic corticosteroids defined as 1-2mg/kg prednisone equivalent daily (either oral or intravenous) with a taper over 4-6 weeks as defined by society consensus guidelines102-105; AND
* No receipt of biologic such as but not limited to (TNFα inhibitor infliximab OR α₄β₇ integrin inhibitor vedolizumab) prior to enrollment.
* Patients must have received steroids to be eligible.
* Steroid "resistant" disease: patients whose symptoms responded (reduction in a CTCAE grade) initially but who developed recurrence upon steroid taper or discontinuation.
* Steroid "refractory" disease: patients whose symptoms have not clinically improved by a CTCAE grade in ≥48 hours or maximum of 14 days.

  * Patient may have received any number of lines of prior systemic therapy.
  * Patient with any solid tumor or hematologic malignancy are eligible.
  * Patient must not be receiving concurrent radiation therapy.
  * Willingness to undergo cohort-specific evaluation.
* Cohort 1: Dermatologic evaluation, and skin biopsy evaluation prior to and after MTP-101-C administration.
* Cohort 2: GI evaluation, and endoscopic evaluation including colonoscopies prior to and after MTP-101-C administration.

  * Willingness to undergo correlative blood and stool sampling.
  * Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2.
* Patients with ECOG PS 2 wherein the decline in PS from baseline is deemed secondary to IMC may be enrolled at the discretion of Sponsor-Investigator.
* Patients with ECOG PS 2 wherein PS is at baseline and deemed secondary to disease are excluded.

  * Have adequate organ function per specimens must be collected within 7 days prior to the start of study treatment.

Exclusion Criteria:

* Multiple irAEs besides irCAE or IMC.

  * Patients with concurrent ≥Grade 3 irAEs besides irCAE or IMC that necessitate systemic immune suppression are not candidates for this trial.
  * Patients with irCAE and/or IMC that are not otherwise clarified in Section 5.1.5 (irCAE including alopecia etc.) are not candidates for this trial.
  * Patients with concomitant irAEs that are well controlled (≤Grade 1 or Grade 2 on repletion medication) may be enrolled at the discretion of Sponsor-Investigator.
* Diagnosis of immunodeficiency, immunosuppression or any other form of immunosuppressive therapy besides steroids/biologics within 7 days prior to the first dose of MTP-101-C treatment.
* Patients at high risk of MDRO colonization including: nursing home residence, age >85, underlying diseases (dementia, poorly controlled diabetes, chronic wounds), in-dwelling medical devices (urinary catheters, feeding tubes, PEG tubes) and a prior history of MDRO colonization.
* Contraindication to endoscopy (cohort 2 only).
* Contraindication to MTP-101-C administration.
* Any prior head/neck and/or abdominal surgery resulting in potentially altered absorption of orally administered FMT pills.
* Active bacterial infection requiring systemic antibiotic therapy.
* Received live vaccines within 30 days prior to the first dose of study treatment and while participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2031-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 2 months
  Incidence of adverse events (AEs) in ICB-treated cancer patients treated with MTP-101-C.
Incidence of Dose-Limiting Toxicities (DLTs) | Up to 2 months
  Incidence of dose-limiting toxicities (DLTs) in ICB-treated cancer patients treated with MTP-101-C. DLT is defined as any adverse event(s) (AEs) considered possibly, probably, or definitely related to MTP-101-C, which occur during the treatment phase. During DLT monitoring period, no further accrual will be permitted. Any patient who has started the studied treatment will be evaluable for safety. AEs will be considered DLTs if deemed related to study therapy: Hematologic: Grade 4 neutropenia, Febrile neutropenia, Grade ≥ 3 neutropenic infection, Grade ≥ 3 thrombocytopenia with bleeding, Grade 4 thrombocytopenia. Non-hematologic: Grade ≥ 3 toxicities (non-laboratory), Grade ≥ 3 nausea, vomiting or diarrhea despite maximal medical intervention, Grade 4 aspartate aminotransferase (AST) and alanine aminotransferase (ALT). Other (non-AST/ALT) non-hematologic Grade ≥ 3 laboratory value if the abnormality leads to overnight hospitalization

SECONDARY OUTCOMES:
Resolution of steroid relapsed/refractory irCAEs (cohort 1) | Up to 2 months
  Resolution of steroid relapsed/refractory irCAEs (cohort 1) following MTP-101-C using cohort -specific endpoints including modified CTCAE grading system (cohort 1)
Resolution of steroid relapsed/refractory IMC (cohort 2) | Up to 2 months
  Resolution of steroid relapsed/refractory IMC (cohort 2) following MTP-101-C using cohort -specific endpoints including modified CTCAE grading system (cohort 1) or endoscopic assessment scale Full Mayo Score (FMS) (cohort 2). FMS includes Partial Mayo Score (PMS) plus endoscopic findings. PMS assesses Stool frequency (per day - normal number of stools to ≥ 5 more, Rectal bleeding (none to blood alone passes) and Physician's global assessment (normal to severe disease), all with scores ranging from 0 to 3. Scores range from 0 - 9 points. Endoscopic score findings range from 0 - 3. Total full scores range from 0 to12, with higher scores indicating more severe ulcerative colitis.
Resolution of IMC following MTP-101-C in steroid relapsed/refractory irCAE (cohort 1) | Up to 2 months
  Resolution of IMC following MTP-101-C in steroid relapsed/refractory irCAE (cohort 1) or IMC (cohort 2) using clinical endpoint Partial Mayo Score (PMS), which assesses Stool frequency (per day - normal number of stools to ≥ 5 more, Rectal bleeding (none to blood alone passes) and Physician's global assessment (normal to severe disease), all with scores ranging from 0 to 3. Scores range from 0 - 9 points, with higher scores indicating more severe ulcerative colitis.
Resolution of IMC following MTP-101-C in steroid relapsed/refractory IMC (cohort 2) | Up to 2 months
  Resolution of IMC following MTP-101-C in steroid relapsed/refractory irCAE (cohort 1) or IMC (cohort 2) using clinical endpoint Partial Mayo Score (PMS), which assesses Stool frequency (per day - normal number of stools to ≥ 5 more, Rectal bleeding (none to blood alone passes) and Physician's global assessment (normal to severe disease), all with scores ranging from 0 to 3. Scores range from 0 - 9 points, with higher scores indicating more severe ulcerative colitis.
Patient Reported Outcomes - FACT-ICM | At Screening, Day +28 through Day +35, Day +42 through Day +49
  The FACT-ICM is a self-administered questionnaire that measures quality of life within the prior 7 days in patients being treated with immunotherapy, using 52 items with a 5-point Likert-type scale, (0 = Not at all to 5 = Very Much). Subscales include Physical Well-Being max score=28), Social/Family Well-Being (max score=28), Emotional Well-Being (max score=24), Functional Well-Being (max score=28), Immune Checkpoint Modulator Subscale (max score=100). Total scores= 0 to 208, with higher scores indicating better quality of life.
Patient Reported Outcomes - FACIT-general | At Screening, Week 1, Week 2, Week 3, Week 4
  FACIT-general is a self-administered questionnaire that measures quality of life within the prior 7 days in patients being treated with immunotherapy, using 27 items with a 5-point Likert-type scale, (0 = Not at all to 5 = Very Much). Subscales include Physical Well-Being max score=28), Social/Family Well-Being (max score=28), Emotional Well-Being (max score=24), Functional Well-Being (max score=28), Total scores= 0 to 108, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Diwakar M Davar, MD, PhD, Principal Investigator — UPMC Hillman Cancer Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No